CLINICAL TRIAL: NCT06760221
Title: Safety and Efficacy of Preoperative Stereotactic Body Radiotherapy (SBRT) and Radical Surgery for Soft Tissue Sarcoma of Extremities
Brief Title: Safety and Efficacy of Preoperative SBRT and Radical Surgery for Soft Tissue Sarcoma of Extremities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0177
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Soft Tissue Sarcoma; Stereotactic Body Radiotherapy; Surgery
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: neoadjuvant stereotactic body radiation therapy followed by radical surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- radiotherapy (Experimental): neoadjuvant stereotactic body radiation therapy followed by radical surgery
  Interventions: Radiation: stereotactic body raiotherapy

INTERVENTIONS:
Radiation: stereotactic body raiotherapy — Neoadjuvant stereotactic body radiation therapy followed by radical surgery for soft tissue sarcoma.

SUMMARY:
Currently, the effectiveness and safety of preoperative hypo-fractionated radiotherapy in treating extremity soft tissue sarcomas remain inconclusive, warranting further investigation. Optimizing the neoadjuvant radiotherapy approach, including fractionation schedules and the interval between radiotherapy and surgery, is crucial to enhancing clinical efficacy while ensuring safety. This study proposes a multicenter, prospective, single-arm clinical trial utilizing preoperative SBRT for patients with high-grade extremity STS, tumors larger than 5 cm, or cases where achieving safe surgical margins is challenging due to involvement of surrounding blood vessels or nerves. The trial aims to preliminarily assess the impact of preoperative SBRT followed by radical surgery on surgical safety, quality of life, and tumor control in these patients.

DETAILED DESCRIPTION:
The effectiveness and safety of preoperative hypo-fractionated radiotherapy in treating extremity soft tissue sarcomas remain inconclusive, warranting further investigation. Optimizing the neoadjuvant radiotherapy approach, including fractionation schedules and the interval between radiotherapy and surgery, is crucial to enhancing clinical efficacy while ensuring safety. This study proposes a multicenter, prospective, single-arm clinical trial utilizing preoperative SBRT for patients with high-grade extremity STS, tumors larger than 5 cm, or cases where achieving safe surgical margins is challenging due to involvement of surrounding blood vessels or nerves. The trial aims to preliminarily assess the impact of preoperative SBRT followed by radical surgery on surgical safety, quality of life, and tumor control in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. Confirmed diagnosis of soft tissue sarcomas;
3. Highly malignant soft tissue sarcomas;
4. Not received surgery, chemotherapy or other antitumor therapy;
5. ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1;
6. Signed informed consent;
7. Willing to provide tissue from an excisional biopsy of a tumor lesion，willing to provide blood sample before and after treatment;

Exclusion Criteria:

1. Patients with soft tissue sarcoma of extremities with shallow tumor location, small size, low grade pathology and operable surgical resection;
2. Distant metastasis;
3. Received surgery or chemotherapy or other antitumor therapy;
4. Previously participated in other clinical trials;
5. History of severe allergies, patients with allergic conditions, such as contrast agent allergy;
6. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
7. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy;
8. Active infection requiring systemic therapy;
9. Known psychiatric or substance abuse disorders ;
10. Pregnant or breastfeeding;
11. Known history of human immunodeficiency virus (HIV: HIV 1/2 antibodies);
12. Received a live vaccine within 30 days before radiotherapy.
13. Unable to lie flat.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of radiotherapy followed by radical surgery | 120 days after radical surgery
  Incidence of Treatment-Emergent Adverse events (CTCAE v5.0)

SECONDARY OUTCOMES:
Extremity function and Quality of life by EORTC QLQ-C30 | Assessed up to 12 months
  1 year after radical surgery
Recurrence free survival | 1-,2-,3-year after radical surgery
  From date of enrollment to the date of first documented recurrence
Progression free survival | 1-,2-,3-year after radical surgery
  from date of enrollment to the date of first documented progression
Overall survival | 1-,2-,3-year after radical surgery
  from date of enrollment to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Qichun Wei, MD/PhD, Principal Investigator — Zhejiang University
Locations (1):
- the second affiliated hospital of Zhejiang University Hangzhou, Zhejiang, China, 310009, Hangzhou, Zhejiang, China